CLINICAL TRIAL: NCT05229627
Title: Multimodal Magnetic Resonance Imaging Study on the Neural Mechanisms of Remission in Children With ADHD Treated With Methylphenidate or Atomoxetine
Brief Title: Multimodal Magnetic Resonance Imaging Study on the Neural Mechanisms of Remission in Children With ADHD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Sixth Hospital (Other)
Collaborators: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Qingjiu Cao, Assoc Prof. Dr., Peking University Sixth Hospital
Other Study IDs: NSFC81471382
Record Dates: First submitted 2015-12-31; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: ADHD
Keywords: multimodule MRI, remission, MPH, ATX, ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- healthy control: healthy controls, screened by K-SADS-PL
- MPH induced Remission: patients show remission after 8-12 weeks of treatment with MPH
  Interventions: Drug: MPH
- non responder to MPH: patients don't show remission after 8-12 weeks of treatment with MPH
  Interventions: Drug: MPH
- ATX induced remission: patients show remission after 8-12 weeks of treatment with ATX
  Interventions: Drug: ATX
- non responder to ATX: patients don't show remission after 8-12 weeks of treatment with ATX
  Interventions: Drug: ATX

INTERVENTIONS:
Drug: MPH — the drug would be prescribed to patients without any contraindication
  Other Names: Concerta
  Groups: MPH induced Remission; non responder to MPH
Drug: ATX — the drug would be prescribed to patients without any contraindication
  Other Names: Strattera
  Groups: ATX induced remission; non responder to ATX

SUMMARY:
Attention-deficit/hyperactivity disorder(ADHD) is highly prevalent among children and adolescents and often associated with poor long-term outcomes in adulthood. it is thus a serious public health problem. Methylphenidate(MPH) and Atomoxetine(ATX) are most frequently used for treating ADHD in many countries but the individual treatment response varies. Some patients present good response to either MPH or ATX with minimal or no symptoms left and optimal functioning(remission) after treatment, while others are poor responders to one of the two or even both. The underlying mechanism for the heterogenous responsiveness remains unknown. Thus we proposed to use multimodule magnetic resonance imaging(MRI) technology to explore the neural mechanisms of remission in children with ADHD treated with MPH or ATX.

DETAILED DESCRIPTION:
the main aim of the current study is to explore the mechanism of remission in children with ADHD treated by MPH or ATX. Baseline information including demographic information, clinical features including ADHD symptoms, cognitive assessments such as executive function, MRI scans including resting state functional MRI, structural MRI, and DTI would be acquired in each participant. after 8-12 weeks of treating with MPH or ATX, patients would be classified into subgroups of remitted and unremitted groups. all baseline tests would be acquired again at the end of the study. comparisons would be done to explore the remission mechanism induced by MPH or ATX

ELIGIBILITY:
Inclusion Criteria:

- clinical diagnosis of ADHD, based on K-SADS-PL medication naive aged 6-16

Exclusion Criteria:

- history of severe head injury (with coma) other severe physical problem or disease in nervous system intelligence quotient (IQ) < 80

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: the ADHD group would be recruited by the clinic for child psychiatry in Peking University sixth hospital; while the healthy control would be recruited in community setting
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Swanson, Nolan and Pelham , Version Ⅳ Rating Scale (SNAP-Ⅳ) | 8 to 12 weeks
  to define remission, using Swanson, Nolan and Pelham , Version Ⅳ Rating Scale (SNAP-Ⅳ), both in baseline and follow-up
Clinical Global Impressions-Improvement scale (CGI-I) | 8 to 12 weeks
  to define remission, participants will assessed by CGI-I in follow-up, and Clinical Global Impressions-Severity scale (CGI-S) in baseline.
resting state functional magnetic resonance imaging (rs-fMRI) | 8 to 12 weeks
  participants undergo resting state functional MRI (rs-fMRI) scan both in baseline and follow-up, and the duration for each rs-fMRI is 8 minutes.
side effect assessment | 8 to 12 weeks
  with clinical global impression scale

SECONDARY OUTCOMES:
Structural magnetic resonance imaging (sMRI) | 8 to 12 week
  participants undergo structural magnetic resonance imaging (sMRI) scan both in baseline and follow-up, and the duration for each sMRI is 5 minutes.
Diffusion Tensor Imaging (DTI) | 8 to 12 weeks
  participants undergo DTI scan both in baseline and follow-up, and the duration for each sMRI is 10 minutes.
WEISS Functional Impairment Rating Scale-parent report (WFIRS-P) | 8 to 12 weeks
  to assess the improvement of social function impairment in ADHD, participants will finish the WFIRS-P both in baseline and follow-up
Behavior Rating Inventory of Executive Function (BRIEF) | 8 to 12 weeks
  to assess the improvement of ecological executive function in ADHD, participants will finish the BRIEF both in baseline and follow-up
The Cambridge Neuropsychological Tests Automated Battery（CANTAB） | 8 to 12 weeks
  to assess the improvement of neuropsychological executive function in ADHD, participants will finish the executive functional test measured by CANTAB both in baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Qingjiu Cao, PhD, Principal Investigator — Peking University Sixth Hospital

IPD SHARING:
Plan to Share IPD: Undecided
the data would be published first and not yet decided to share with other research groups